CLINICAL TRIAL: NCT07219992
Title: Testing a Novel Parent-Based Treatment for Adolescent Anxiety Disorders
Brief Title: Parent-Based Treatment for Adolescent Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: MQ: Transforming Mental Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000040413
Record Dates: First submitted 2025-10-20; First posted 2025-10-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Disorder of Adolescence

STUDY DESIGN:
Masking Description: Adolescent participants and their parents will be enrolled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Parenting for Anxious Childhood Emotions (SPACE) (Experimental): A parent-only approach to treating anxiety disorders in adolescents delivered over 12 sessions.
  Interventions: Behavioral: Supportive Parenting for Anxious Childhood Emotions (SPACE)
- Parent Education and Support (PES) (Active Comparator): Parent-based approach comparator arm delivered over 12 sessions.
  Interventions: Behavioral: Parent Educational Support (PES)

INTERVENTIONS:
Behavioral: Supportive Parenting for Anxious Childhood Emotions (SPACE) — Parent based treatment delivered by a therapist 12 weekly sessions with parents.
  Arms: Supportive Parenting for Anxious Childhood Emotions (SPACE)
Behavioral: Parent Educational Support (PES) — Parent Educational Support: 12 weekly sessions with parents
  Arms: Parent Education and Support (PES)

SUMMARY:
This study aims to test the efficacy of a parent-only approach to treating anxiety disorders in adolescents: SPACE (Supportive Parenting for Anxious Childhood Emotions). The comparator is another parent-based approach, PES (Parent Education and Support). The study design is a randomized controlled trial with 2 treatment arms and 3 assessment points (pre, post, and follow-up) using questionnaire data and clinical interviews.

DETAILED DESCRIPTION:
The primary objective is to examine if SPACE is more efficacious than PES in reducing adolescent anxiety symptoms. The secondary objective is to examine if SPACE produces greater change than PES in improving family accommodation and family functioning.

SPACE and PES will be delivered over 12 sessions: Sessions 1-6 (once weekly), a mid-treatment assessment, Sessions 7-12 (once weekly), and a Post-treatment assessment.

Sessions can be attended in person or via Zoom.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for a primary DSM-5 AD, including separation anxiety disorder, social anxiety disorder, generalized anxiety disorder, specific phobia, panic disorder, and agoraphobia (determined by the ADIS-C/P).
* Cease all other psychosocial treatment, upon consultation with the project staff and service provider.
* Not currently use any psychotropic medication, other than a stable dose (i.e., same dose for a minimum of 6 months prior to enrollment; no changes during course of the study) of a stimulant medication or selective serotonin reuptake inhibitor (SSRI).
* Have an eligible and willing participating parent (see parent exclusions below).

Exclusion Criteria:

Adolescent:

* Meet criteria for any DSM-5 disorder more impairing than the most impairing AD (determined by the ADIS-C/P).
* Have any of the following disorders: autism spectrum disorder; intellectual disability; neurocognitive disorders; bipolar disorder; schizophrenia and other psychotic disorders; and alcohol and substance use disorders (determined by the Health History Form and ADIS-C/P).
* Report a suicide attempt in the last 3 months, or current suicide intent and plans (determined by the ASQ).
* Be a victim of past or present undisclosed abuse requiring investigation or ongoing supervision by the Department of Social Services.
* Not have sufficient proficiency with the English language to complete assessments.

Parents:

* Have any of the following: intellectual disability; neurocognitive disorders; untreated bipolar disorder; untreated schizophrenia and other psychotic disorders; and untreated alcohol and substance use disorders (determined by the Health History Form).
* Not be living with the adolescent at least 50% of the time for at least one year prior to enrollment.
* Not have sufficient proficiency with the English language to complete assessments and treatment.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Mean Pediatric Anxiety Rating Scale (PARS) score | Week 1 and 14
  This scale measures anxiety symptoms on 7 dimensions (e.g., avoidance, severity) from 0 ("minimal") to 5 ("extreme"). Total scores range from 0 - 35. Higher scores indicate greater anxiety severity.
Mean Screen for Child Anxiety Related Emotional Disorders (SCARED-C/P) score | Week 1, 7 and 14
  This scale assesses adolescent anxiety symptoms on a 3-point scale (0 "not true/hardly ever true" to 2 "very true/often true") with total score range = 0 - 82. Higher scores suggest greater anxiety symptoms.
Mean Child Anxiety Impact Scale (CAIS-C/P) score | Week 1 and 14
  This scale assesses adolescent anxiety that specifically captures impairment related to anxiety across important domains of functioning. Adolescents and parents rate items on a 4-point scale (0 "not at all" to 3 "very much"); total score range = 0 - 81. Higher scores suggest greater anxiety symptoms.
Clinical Global Impression Scale - Severity (CGI-S) and Improvement (CGI-I) scales score | Week 1 and 14
  This measure will be used to assess overall severity (CGI-S) and improvement (CGI-I) in adolescent anxiety. Total score range for each is 1-7. (Scores of 1 ("very much improved/normal") or 2 ("much improved/borderline ill") indicate a positive treatment response; all other responses are considered negative responses. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Mean Family Accommodation Scale - Anxiety (FASA-C/P) score | Week 1, 8 and 14
  This scale assesses family accommodation. Adolescents and parents rate 9 items on a 5-point scale, 0 "never" to 4 "daily"; total score range = 0 - 36. Higher scores indicate more accommodation.
Mean Family Assessment Device - General Functioning Scale (FAD-GF) score | Week 1 and 14
  This scale will measure of overall family functioning. Adolescents and parents rate 12-items on a 4-point scale (0 "strongly disagree" - 3 "strongly agree"). Total score range 0-3. Higher scores indicate more unhealthy family functioning.
Mean Parent Problem Checklist scale score | Week 1 and 14
  This scale will measure co-parenting and assesses parents' ability to cooperate and work together in family management. Parents rate 16 items on a yes/no scale to form the Overall Problems scale, total score range = 0 - 16. Higher scores indicate greater conflict. Parents also rate each "yes" on a 7-point scale (1 "not at all" to 7 "very much") to form the Extent scale. Total score range 16-112. Higher scores indicate greater extent of a problem for them and their partner.
Mean Parent Behavior Inventory - Child and Parent Report (CRPBI/PRPBI) scale score | Week 1 and 14
  This scale will measure parent-child relationship quality. Adolescents and parents respectively rate 30-items assessing perceived parental behaviors on a scale from 0 ("Not like") to 2 ("A lot like"). Total score range = 0 to 2 with higher scores indicating better relationship quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Etkin, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No